CLINICAL TRIAL: NCT00106119
Title: Peripheral Thyroid Hormone Conversion and Glucose and Energy Metabolism
Brief Title: Thyroid and Glucose and Energy Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kong Chen, Ph.D., Clinical Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 050119; 05-DK-0119 (Other: NIH)
Record Dates: First submitted 2005-03-19; First posted 2005-03-21 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Thyroid Diseases
Keywords: Levothyroxine; Liothyronine; Lipid Metabolism; Gluconeogensis; Thyrotropin Releasing Hormone; Deiodinase; Replacement Thyroid Hormone Therapy; Thyroidectomy; Near Total Thyroidectomy
MeSH Terms: conditions — Thyroid Diseases | interventions — Triiodothyronine; Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liothyronine and Levothyroxine (Active Comparator): Hypothyroid patients treatment with Levothyroxine and Liothyronine in 2 crossover, randomized phases
  Interventions: Drug: Liothyronine and Levothyroxine

INTERVENTIONS:
Drug: Liothyronine and Levothyroxine — Hypothyroid patients are treated with Liothyronine and Levothyroxine in 2 crossover, randomized phases
  Other Names: T3 and T4

SUMMARY:
This study will examine how two thyroid preparations-levothyroxine (T4) and liothyronine (T3)-affect fat and cholesterol metabolism, blood sugar regulation, and thyrotropin secretion in patients who have had their thyroid gland removed. Results of the study may help in the development of better therapies to optimize blood sugar and cholesterol levels in some patients.

Patients 18 years of age or older who have had most or all of their thyroid gland removed and are taking long-term thyroid hormone medication may be eligible for this study after screening.

DETAILED DESCRIPTION:
Thyroid hormone action plays an important role in the regulation of many physiologic processes, among them glucose and lipid metabolism. Interestingly, the clinical presentation of thyroid dysfunction is extremely variable, with relatively poor correlation between circulating hormone levels and clinical features. This finding suggests that the local, intracellular concentration of the active hormone liothyronine (T3), regulated by peripheral conversion of the pro-hormone levothyroxine (T4), is an important determinant in the maintenance of the thyroidal homeostasis.

The aim of the present study is the evaluation of the role of peripheral thyroid hormone conversion in the regulation of glucose and lipid metabolism by assessing the differential response to T4 or T3 treatment in subjects devoid of endogenous thyroid hormone production. T3 administration bypasses peripheral metabolism and therefore will allow us to assess the role of the peripheral thyroid hormone conversion in the regulation of the hormone action at the end-organ level.

Fifty hypothyroid subjects will be initially randomized to either of the thyroid hormone replacements liothyronine (T3) or levothyroxine (T4) treatment period (one arm cross-over design, with treatment sequence randomized), aimed to maintain serum TSH levels greater than or equal to 0.5 less than or equal to 1.5 mU/L, indicating full replacement. After a 30-day period of steady-state replacement the study subjects will be admitted to the Clinical Center and, after a three-day period of stabilization and an overnight fast, will undergo the following tests: escalating dose TRH stimulation test, indirect calorimetry, graded exercise tolerance test, DEXA scan, and echocardiogram.

Patients will also undergo skeletal muscle biopsy and subcutaneous adipose tissue biopsy and microdialysis, as well as a two-step euglycemic hyperinsulinemic clamp with measurement of splanchnic gluconeogenesis. Fasting venous blood samples will be collected for the determination of the parameters of lipid, glucose and energy metabolism.

After discharge, the patients will switch to the other form of thyroid hormone replacement therapy (second period) . The therapy will be adjusted in order to achieve the same therapeutic goal for TSH concentrations (greater than or equal to 0.5 less than or equal to 1.5 mU/L), analogous to that achieved during the first phase of the study (TSH less than or equal to 0.5 mU/L difference between T3 and T4 phases). After reaching a 30-day period of steady-state replacement, study subjects will be re-admitted to the Clinical Center and the previously described evaluation procedures will be repeated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years, male or female.

History of total or near total thyroidectomy or hypothyroidism on replacement therapy.

For non-thyroidectomized patients, at least three-year history of replacement therapy (at least 1.2 mcg/Kg LT4/body weight), and less than 5% uptake at 24H on (123)I thyroid scan while on replacement therapy.

Written informed consent.

EXCLUSION CRITERIA:

BMI less than or equal to 20 or greater than or equal to 30 kg/m(2).

Metastatic thyroid cancer or history of thyroid cancer with high risk of recurrence requiring suppressive thyroid hormone therapy (Singer 1996).

Significant thyroid residual greater than 1 mL as measured by ultrasound (limited to thyroidectomized patients) or greater than 5 percent uptake at 24H on (123)I thyroid scan while on replacement therapy (limited to hypothyroid patients not undergone total thyroidectomy).

History or symptoms compatible with cardiovascular disease, including paroxysmal supraventricular tachycardia, atrial fibrillation, syncopal episodes or use of prescription medications for heart conditions, including antihypertensives.

Allergy to lidocaine, isoproterenol, TRH, levothyroxine, liothyronine, Tylenol #3, oxycodone, nitroglycerin.

Pregnancy or unwillingness to use non-hormonal contraception during the study.

Breastfeeding

Use of hormonal contraceptives or estrogen replacement therapy.

Use of tobacco (smoking, chewing) for the two weeks preceding the hospital admissions (metabolic testing)

Diabetes mellitus, either type I or II.

Hypercholesterolemia (serum levels greater than or equal to 240 mg/dL), hypertriglyceridemia (plasma levels greater than or equal to 220 mg/dL) and/or use of antilipemic therapy.

Liver disease or ALT serum level greater than two fold the upper laboratory reference limit.

Renal insufficiency or estimated creatinine clearance less than or equal to 50 mL/min.

Use of medications/supplements/alternative therapies known to alter thyroid function.

Current history or symptoms compatible with psychosis including major depression (including history of hospitalization for depression, history of attempted suicide, history of suicidal ideation).

Use of antipsychotic medications

History of drug or alcohol abuse within the last 5 years; current use of drugs or alcohol (CAGE greater than 3).

Keloid formation (relative to skeletal muscle and subcutaneous adipose tissue biopsies).

Current or previous clinically significant (requiring medical/surgical intervention) extrathyroidal manifestations of autoimmune thyroid disease (dermopathy, ophthalmopathy, arthropathy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arner P, Bolinder J, Wennlund A, Ostman J. Influence of thyroid hormone level on insulin action in human adipose tissue. Diabetes. 1984 Apr;33(4):369-75. doi: 10.2337/diab.33.4.369. PMID 6423430
- [Background] Bakker SJ, ter Maaten JC, Popp-Snijders C, Slaets JP, Heine RJ, Gans RO. The relationship between thyrotropin and low density lipoprotein cholesterol is modified by insulin sensitivity in healthy euthyroid subjects. J Clin Endocrinol Metab. 2001 Mar;86(3):1206-11. doi: 10.1210/jcem.86.3.7324. PMID 11238510
- [Background] Bartha T, Kim SW, Salvatore D, Gereben B, Tu HM, Harney JW, Rudas P, Larsen PR. Characterization of the 5'-flanking and 5'-untranslated regions of the cyclic adenosine 3',5'-monophosphate-responsive human type 2 iodothyronine deiodinase gene. Endocrinology. 2000 Jan;141(1):229-37. doi: 10.1210/endo.141.1.7282. PMID 10614643
- [Derived] Yavuz S, Linderman JD, Smith S, Zhao X, Pucino F, Celi FS. The dynamic pituitary response to escalating-dose TRH stimulation test in hypothyroid patients treated with liothyronine or levothyroxine replacement therapy. J Clin Endocrinol Metab. 2013 May;98(5):E862-6. doi: 10.1210/jc.2012-4196. Epub 2013 Apr 12. PMID 23585666
- [Derived] Celi FS, Zemskova M, Linderman JD, Smith S, Drinkard B, Sachdev V, Skarulis MC, Kozlosky M, Csako G, Costello R, Pucino F. Metabolic effects of liothyronine therapy in hypothyroidism: a randomized, double-blind, crossover trial of liothyronine versus levothyroxine. J Clin Endocrinol Metab. 2011 Nov;96(11):3466-74. doi: 10.1210/jc.2011-1329. Epub 2011 Aug 24. PMID 21865366
- [Derived] Celi FS, Zemskova M, Linderman JD, Babar NI, Skarulis MC, Csako G, Wesley R, Costello R, Penzak SR, Pucino F. The pharmacodynamic equivalence of levothyroxine and liothyronine: a randomized, double blind, cross-over study in thyroidectomized patients. Clin Endocrinol (Oxf). 2010 May;72(5):709-15. doi: 10.1111/j.1365-2265.2009.03700.x. PMID 20447070
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-DK-0119.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from NIH Clinical Center, Bethesda, Maryland, USA between June 2005 and November 2007.
Pre-assignment Details: 110 participants inquired through phone; 24 screened, 10 excluded 8 did not meet inclusion criteria and 2 refused participation).
Groups:
- Liothyronine First, Then Levothyroxine: Liothyronine (dose of 2.5, 10, or 16 mcg) in first intervention period and Levothyroxine (dose of 5, 10, or 33 mcg) in second intervention period (after washout period)
- Levothyroxine First, Then Liothyronine: Levothyroxine (dose of 5, 10, or 33 mcg) in first intervention period and Liothyronine (dose of 2.5, 10, or 16 mcg) in second intervention period (after washout period)
Period: First Intervention
Arm/Group | Liothyronine First, Then Levothyroxine | Levothyroxine First, Then Liothyronine
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout Period of 30 Days
Arm/Group | Liothyronine First, Then Levothyroxine | Levothyroxine First, Then Liothyronine
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Liothyronine First, Then Levothyroxine | Levothyroxine First, Then Liothyronine
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who completed the study
Groups:
- Entire Study Population: Includes groups randomized to receive Levothyroxine first and Liothyronine first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 14
Duration of hypothyroidism [Mean (Standard Deviation); unit: years] | 8.6 (13.1)
Thyroid stimulating hormone (TSH) [Mean (Standard Deviation); unit: mU/liter] | 1.1 (1.4)
Triiodothyronine (T3) [Mean (Standard Deviation); unit: ng/dl] | 99.0 (24.2)
Free thyroxine (T4) [Mean (Standard Deviation); unit: ng/dl] | 1.76 (0.46)

OUTCOME MEASURES:

1. Primary Outcome: Insulin-mediated Glucose Disposal Rate at Levothyroxine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Groups:
- Liothyronine/Levothyroxine Therapy Intervention Arm: Hypothyroid patients are treated with Levothyroxine and Liothyronine in 2 crossover, randomized phases
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/kg/min | 7.26 (2.7)

2. Secondary Outcome: Total Cholesterol at Levothyroxine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 196 (26)

3. Primary Outcome: Insulin-mediated Glucose Disposal Rate at Liothyronine Treatment Phase
Time Frame: One month of therapy
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/kg/min | 7.37 (4.4)

4. Secondary Outcome: Total Cholesterol at Liothyronine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 174 (28)

5. Secondary Outcome: Triglycerides at Levothyroxine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 152 (31)

6. Secondary Outcome: Triglycerides at Liothyronine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 144 (16)

7. Secondary Outcome: Resting Energy Expenditure at Levothyroxine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: kcal/24 hour
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
kcal/24 hour | 1201 (282)

8. Secondary Outcome: Resting Energy Expenditure at Liothyronine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: kcal/24 hour
Groups:
- Liothyronine/Levothyroxine Therapy Intervention ArmArm: Hypothyroid patients are treated with Levothyroxine and Liothyronine in 2 crossover, randomized phases
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention ArmArm
Number analyzed (Participants) | 14
kcal/24 hour | 1177 (323)

9. Secondary Outcome: Left Ventricle Mass Index at Levothyroxine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
g/m^2 | 71 (16)

10. Secondary Outcome: Left Ventricle Mass Index at Liothyronine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
g/m^2 | 71 (19)

11. Secondary Outcome: Apolipoprotein A-I at Levothyroxine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 152 (31)

12. Secondary Outcome: Apolipoprotein A-I at Liothyronine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 144 (16)

13. Secondary Outcome: Apolipoprotein B at Levothyroxine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 87 (19)

14. Secondary Outcome: Apolipoprotein B at Liothyronine Treatment Phase
Time Frame: One month of therapy.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Liothyronine/Levothyroxine Therapy Intervention Arm
Number analyzed (Participants) | 14
mg/dl | 72 (15)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Levothyroxine Period: Patients at Levothyroxine Period
- Liothyronine Period: Patients at Liothyronine Period
Arm/Group | Levothyroxine Period | Liothyronine Period
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine Period (N=14) | Liothyronine Period (N=14)
General disorders (General disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine Period (N=14) | Liothyronine Period (N=14)
generalized anxiety disorder (Psychiatric disorders) | 1 (14) | 0 (0) — This adverse event could not be separated between two treatment periods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes